CLINICAL TRIAL: NCT05252585
Title: Phase IV, Prospective Single Arm Study of Safety and Efficacy of Votubia (Everolimus) in Taiwanese Adults With Tuberous Sclerosis Complex Who Have Renal Angiomyolipoma
Brief Title: A Phase IV Study of Safety and Efficacy of Everolimus in Taiwanese Patients With Tuberous Sclerosis Complex Who Have Renal Angiomyolipoma (TSC-AML)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001M2402
Record Dates: First submitted 2022-02-16; First posted 2022-02-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Renal Angiomyolipoma
Keywords: Tuberous Sclerosis Complex; TSC; Angiomyolipoma; AML; Everolimus
MeSH Terms: conditions — Angiomyolipoma; Tuberous Sclerosis | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Everolimus (Experimental): Participants with confirmed diagnosis of TSC-AML and who fulfil the local (Taiwan) reimbursement criteria of everolimus for TSC-AML treatment
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus tablets for oral use. The recommended everolimus starting dose will be 10 mg orally taken once daily for all patients, except for those with impaired liver function, for whom the everolimus dose will be:
  * Child-Pugh grade A: 7.5 mg once daily (for patients with mild hepatic impairment)
  * Child-Pugh grade B: 5.0 mg once daily (for patients with moderate hepatic impairment)
  Other Names: RAD001

SUMMARY:
The purpose of this prospective study is to assess the safety and efficacy of everolimus in Taiwanese patients with renal angiomyolipoma (AML) associated with tuberous sclerosis complex (TSC) . Only patients who fulfil the local reimbursement criteria of everolimus for TSC-AML will be included in this study.

DETAILED DESCRIPTION:
This open-label, prospective, single-arm, multicenter Phase IV post approval commitment (PAC) study is planned to be conducted in approximately 10 patients with confirmed diagnosis of TSC-AML and who fulfil the local reimbursement criteria of everolimus for TSC-AML treatment.

The study will have a 30-day screening phase, and each patient will be on treatment up to 52 weeks. Enrollment will end at the latest within 52 weeks from Day 1 of the study, regardless of the number of patients actually recruited. After completion of the treatment phase/end of treatment (EOT), eligible patients will enter a 4-week safety follow up (FU) phase. Patients who continue to be on treatment beyond 52 weeks, based on the investigator's judgment will not be included in the 4-week safety FU phase.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female patients from ≥ 18 years of age.
2. Signed informed consent must be obtained prior to participation in the study.
3. Participants with TSC associated with renal AML which is eligible for treatment with everolimus per local reimbursement criteria.

Exclusion Criteria:

1. Patients with severe hepatic impairment (Child-Pugh class C)
2. Any severe and/or uncontrolled medical conditions.
3. Pregnant or breast-feeding females.
4. Patients with hypersensitivity to the active substance, to other rapamycin derivatives, or to any of the excipients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-11-25 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with adverse events (AEs), Serious AEs (SAEs) and AEs of special interest (AESI) | From first dose of study treatment up to 56 weeks
  Percentage of participants with AEs, SAEs and AESIs.

SECONDARY OUTCOMES:
Angiomyolipoma (AML) response rate | Up to 52 weeks
  AML response rate is defined as the percentage of patients with an AML response. AML response will be defined as: A reduction in AML volume of at least 50% relative to screening, where AML volume is the sum of the volumes of all target AML identified at screening. In addition, AML response have to satisfy: no new AML ≥ 1 cm in longest diameter are identified, neither kidney increases in volume by more than 20% from nadir (where nadir is the lowest kidney volume at the screening), the participant does not have any angiomyolipoma-related bleeding of grade equal or over 2 (as defined by NCI CTCAE, version 5).
AML progression rate | Up to 52 weeks
  AML progression rate is defined as the percentage of patients with an AML progression. AML progression status is defined as one or more of the following: an increase from nadir of 25% or more in AML volume to a value greater than screening AML (where nadir is the lowest AML volume obtained for the participant previously in the trial), the appearance of a new AML ≥ 1.0 cm in longest diameter, an increase from nadir of 20% or more in the volume of either kidney to a value greater than screening (where nadir is the lowest kidney volume obtained for the participant previously in the trial), angiomyolipoma-related bleeding grade ≥2 (as defined by NCI CTCAE, version 5)
Percentage of participants with laboratory abnormalities | From screening up to 56 weeks
  The laboratory assessment (including hematology, coagulation, biochemistry, and urinalysis) will be recorded at baseline and during the study based on changes in grade of laboratory abnormality.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Taiwan (4):
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Taoyuan District, Taiwan ROC
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com